CLINICAL TRIAL: NCT05637060
Title: A Single Center, Open Label, Randomized, Single-dose, 2 Way Cross-over Study to Explore the Bioequivalence of Vaptor 20mg (Rosuvastatin) Tablet and Crestor 20mg (Rosuvastatin) Tablet Under Fasting Conditions in Healthy Male Pakistani Subjects
Brief Title: Bioequivalence Study of Rosuvastatin Tablet
Acronym: BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: The Searle Company Limited (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-027-ROS-2018/Protocol/1.0
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy Individuals
Keywords: Bioequivalence Study
MeSH Terms: interventions — Drug Evaluation; Tablets; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: A single center, open label, randomized, single-dose, two period, two-way, cross-over study. Subjects will receive one single dose per treatment period separated by a wash-out period of 7 days.
Masking Description: Only Analysts will be kept blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Subjects will take their assigned study medication (Vaptor 20mg), after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time. Those subjects who received Test Drug in first period will receive Reference drug in 2nd period of the study.
  Interventions: Drug: Test Drug; Drug: Reference Drug
- Reference Group (Active Comparator): Subjects will take their assigned study medication (Crestor 20mg), after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time. Those subjects who received Reference Drug in first period will receive Test drug in 2nd period of the study.
  Interventions: Drug: Test Drug; Drug: Reference Drug

INTERVENTIONS:
Drug: Test Drug — One single dose of Vaptor 20 mg will be administered to subjects after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time.
  Other Names: Vaptor 20 mg Tablet
Drug: Reference Drug — One single dose of Crestor 20 mg will be administered to subjects after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time.
  Other Names: Crestor 20 mg Tablet

SUMMARY:
This study is designed to explore the bioequivalence of Test Product Vaptor (Rosuvastatin) 20 mg Tablet with the reference product Crestor (Rosuvastatin) 20 mg tablet under fasting conditions in healthy Pakistani male subjects.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, single-dose, two-period, two-way, cross-over study. Subjects will receive one single dose per treatment period of Test and Reference Drugs separated by a wash-out period of 7 days. Blood samples will be taken up to 72 hours post-dose. The primary pharmacokinetic parameters will be compared for both drugs to assess the bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 years inclusive.
* Subjects with a body mass index from 18.5 to 30 kg/m2 (both inclusive).
* Subjects who are healthy as determined by routine physical examination, including vital sign monitoring (ie, blood pressure, heart rate, and temperature), 12 Lead ECG, and laboratory analysis (ie, hematology, blood biochemistry, and urinalysis)and viral serology as determined by the investigator.
* Subjects should have a negative urine test for drugs of abuse (MOP (morphine) and THC (tetrahydrocannabinol) will be tested) and alcohol breath analysis at screening and prior to each check-in.
* Subjects will be able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study check-In day.

Exclusion Criteria:

* History of smoking (≥3 cigarettes/day), alcoholism, and test for a drug of abuse, heavy pan or gutka user as judged by teeth/mouth inspection.
* Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
* Subject is allergic to Rosuvastatin and/or other HMG-COA inhibitors.
* Subject has received any investigational drug within 30 days.
* Subjects with salt imbalance in the blood (especially low levels of potassium or magnesium in the blood).
* Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
* Ingestion of OTC drug, within 7 days of drug administration.
* History of intake of any prescribed medicine during a period of 30 days, prior to drug administration day of study.
* History of any significant illness in the last four weeks.
* Subjects with a history of renal impairment, liver disease, hypothyroidism, myopathy and rhabdomyolysis.
* Subject taking any vitamins or herbal supplements within the last 14 days of drug administration.
* Subjects who smoke and/or take nicotine in any form. Non-smoking subjects, who have previously smoked, should at least be non-smoking for 6 months prior to dosing.
* Concomitant treatment with cyclosporine, gemfibrozil, Protease Inhibitors (atazanavir and ritonavir, lopinavir and ritonavir or simeprevir), Coumarin Anticoagulant (warfarin), Niacin, Fenofibrate, Colchicine, ezetimibe, erythromycin, an oral contraceptive/ hormone replacement therapy(Ethinyl estradiol and norgestrel), fusidic acid.
* Consumption of grapefruit and/or its products within 14 days prior to the start of study.
* Subjects who test positive for syphilis (VDRL) or who are known to have serum hepatitis or who are carriers of the Hepatitis B surface antigen (HBsAg) or are carriers of antibodies to hepatitis C virus (anti-HCV) or to the human immunodeficiency virus (HIV-1 or HIV-2).
* Individuals having undergone any major surgery within 3 months prior to the start of the study, unless deemed eligible, otherwise by the Principal Investigator or whomever he may designate.
* Inability to take oral medication.
* Subjects with any condition, which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism, or elimination of drugs.
* Subjects with clinically significant abnormalities in investigations (safety assessments) as determined by the Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration | up to 72 hours post dose
  maximum drug concentration in plasma after dose
Time to reach maximum plasma concentration | 0 to 72 hours post dose
  Time required for the drug to reach maximum plasma concentration
AUC (Area under concentration vs time curve) | 0-72 hours
  Area under the time versus plasma drug concentration curve

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Raza Shah, PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi, Pakistan; Naghma Hashmi (Co-PI), PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi, Pakistan
Locations (1):
- Muhammad Raza Shah, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) can be available upon proper request to the Sponsor.
Supporting Information: CSR